CLINICAL TRIAL: NCT04345510
Title: Testing for COVID-19 Infection in Asymptomatic Persons
Status: Completed | Type: Observational
Sponsor: German Cancer Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: COVID-19-1.0-DKFZ
Record Dates: First submitted 2020-04-12; First posted 2020-04-14 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: COVID-19 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intensive action has been taken around the globe to fight the corona virus SARS-COV-2 (COVID-19) pandemia. Clinical symptoms of the infection appear to be variable, from basically asymptomatic infections and mild, flu-like symptoms up to severe respiratory insufficiency, requiring mechanical ventilation at the intensive care unit, and death. Broad testing for COVID-19 infection has been proven difficult in clinical practice and hampered by limited resources. Urgently needed epidemiological data on the rate of silent, asymptomatic infections in the population and the percentage of individuals that have already developed immunity are still missing. Within this study we therefore plan to (i) determine the proportion of asymptomatic COVID-19 virus carriers in (a) German Cancer Research Center (DKFZ) employees, who work and are present at the center during the time of extended minimum operation and (b) in all DKFZ employees before onboarding when extended minimum operation has been terminated. We plan to (ii) develop a high-throughput assay for COVID-19 testing as well as (iii) a serum-based COVID-19 antibody assay. Finally, we will (iv) analyze for a possible correlation between oral microbiome and COVID-19 infection status.

ELIGIBILITY:
Inclusion Criteria:

DKFZ employee

Exclusion Criteria:

Non DKFZ employee

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: DKFZ employees
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
COVID-19 infection | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- German Cancer Research Center, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No